CLINICAL TRIAL: NCT05414864
Title: Insomnia Prevalence and Treatment Impact on Systemic Hypertension
Acronym: Print-HAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Takeda suspended financial support. The first phase (observational study) is ongoing.
Sponsor: University of Sao Paulo (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Luciano F Drager, MD, PhD, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 5276/21/051
Record Dates: First submitted 2022-05-05; First posted 2022-06-10 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-07

CONDITIONS: Insomnia; Hypertension
Keywords: insomnia; hypertension; Ramelteon; sleep hygiene
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hypertension; Sleep Hygiene | interventions — ramelteon

STUDY DESIGN:
Masking Description: team that evaluate the results of complementary exams
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Other): Sleep hygiene alone (control group)
  Interventions: Behavioral: sleep hygiene
- Intervention Group (Other): Sleep Hygiene and Ramelteone (RozeremTM) 8 mg at night
  Interventions: Drug: Ramelteon (RozeremR); Behavioral: sleep hygiene

INTERVENTIONS:
Drug: Ramelteon (RozeremR) — 8mg daily
  Arms: Intervention Group
Behavioral: sleep hygiene — sleep behavioral guidelines

SUMMARY:
Insomnia is defined as some difficulty in sleep onset, consolidation, duration, or quality, despite appropriate opportunities for getting sleep. In the last decade, there is growing evidence associating insomnia and high blood pressure, (HBP), coronary disease, heart failure, atrial fibrillation, as well as with an increased mortality rate. Despite the previously mentioned advances, the real impact of insomnia on HBP is unknown. It is unclear whether the diagnosis and pharmacologic treatment of insomnia will have an impact on 24-h BP. The aim of this study is to outline the prevalence of insomnia in patients with HBP followed in the ambulatories from the Hypertension Units at InCor and Hospital das Clínicas. The main hypothesis is that the prevalence of insomnia is high and most patients remain undiagnosed and consequently untreated. For this phase, up to 1,500 patients with HBP will be selected. Besides the medical records with demographic and anthropometric data, personal and familiar background, as well as regular medication, all patients will perform three systematic and standardized blood pressure checks on electric monitors.

DETAILED DESCRIPTION:
Prevalence of insomnia in patients with HBP The aim of this study is to outline the prevalence of insomnia in patients with HBP followed by the outpatients' clinics at the InCor and Hospital das Clínicas. The main hypothesis is that the prevalence of insomnia is high and most patients remain undiagnosed and consequently untreated. For this phase, up to 1,500 patients with HBP will be recruited. Besides the medical records with demographic and anthropometric data, personal and familiar background, as well as regular medication, all patients will perform three systematic and standardized blood pressure checks on electric monitors. The average of the second and third checks will be the final result.

Furthermore, the following exams will be made:

1. Definition of the presence of insomnia following the criteria from DSM V and filling up the insomnia severity index.
2. Evaluation of the Pittsburgh Sleep Quality Index.
3. Evaluation of obstructive sleep apnea by NoSAS score.
4. Evaluation of daytime sleepiness by the Epworth Sleepiness Scale.
5. Filling the DDAS form for evaluation of perception and impact of insomnia on the life of HBP patients.
6. Filling the Beck form for depression evaluation.

The clinical characteristics of HBP patients with and without insomnia will be compared testing the hypothesis that patients with insomnia will be under more blood pressure medications and/or uncontrolled bllod pressure than patients without insomnia. If positive, a multivariate analysis will be performed for adjusting for counfonding factors.

ELIGIBILITY:
Inclusion criteria:

* BMI <40Kg/m2;
* Availability to participate
* History of HBP under regular treatment (systolic pressure between 130-160 and diastolic pressure between 80-100 mmHg).

Exclusion criteria:

* Use of benzodiazepines or "Z" drugs;
* Night workers;
* History of severe chronic obstructive pulmonary disease (COPD);
* Heart failure (ejection fraction <40% on echocardiogram);
* Prior stroke;
* Generalized anxiety disorder (GAD-7 >14 points) and severe depression (Beck);
* Severe liver disease;
* Alcohol abuse;
* Advanced chronic kidney disease 4 or 5 (glomerular filtration rate <30ml/min/1.73m2);
* Patient who is on loop diuretics;
* Patient with type 1 diabetes;
* Patient with decompensated type 2 diabetes (Glycated hemoglobin >8%);
* Urinuria Incontinence;
* Prostatism;
* History of active cancer;
* Pregnancy;
* Complex sleep behaviors, suicidal behavior;
* Other formal labeled contraindications, including a history of angioedema with ramelteone and patients using fluvoxamine (a strong inhibitor of CYP1A2)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of insomnia treatment on blood pressure (evaluated by Ambulatory blood pressure monitoring) | 3 months
  To assess the impact of treatment of early insomnia with ramelteon on daytime and nighttime blood presure (in mmHg) in hypertensive patients on 24-hour evaluation of ambulatory blood pressure monitoring.

SECONDARY OUTCOMES:
Efficacy of insomnia treatment on blood pressure (evaluated by office blood pressure) | 3 months
  To evaluate the impact of treating initial insomnia with ramelteone on office blood pressure in hypertensive patients on office blood pressure (in mmHg)
Efficacy of insomnia treatment on Sleep duration | 3 months
  To assess the impact of treating insomnia with ramelteon in hypertensive patients on sleep duration evaluated by actigraphy (and reported in minutes of sleep);
Efficacy of insomnia treatment on sleep quality | 3 months
  To evaluate the impact of treating insomnia with ramelteon in hypertensive patients on sleep quality;
Efficacy of insomnia treatment on subgroups of patients (intending to be a sub-study) | 3 months
  Assess whether the pressure response of insomnia treatment on the primary and secondary outcomes is mediated by the presence of obstructive sleep apnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Schutte-Rodin S, Broch L, Buysse D, Dorsey C, Sateia M. Clinical guideline for the evaluation and management of chronic insomnia in adults. J Clin Sleep Med. 2008 Oct 15;4(5):487-504. PMID 18853708
- [Background] Ford ES, Cunningham TJ, Giles WH, Croft JB. Trends in insomnia and excessive daytime sleepiness among U.S. adults from 2002 to 2012. Sleep Med. 2015 Mar;16(3):372-8. doi: 10.1016/j.sleep.2014.12.008. Epub 2015 Jan 14. PMID 25747141
- [Background] Roth T, Coulouvrat C, Hajak G, Lakoma MD, Sampson NA, Shahly V, Shillington AC, Stephenson JJ, Walsh JK, Kessler RC. Prevalence and perceived health associated with insomnia based on DSM-IV-TR; International Statistical Classification of Diseases and Related Health Problems, Tenth Revision; and Research Diagnostic Criteria/International Classification of Sleep Disorders, Second Edition criteria: results from the America Insomnia Survey. Biol Psychiatry. 2011 Mar 15;69(6):592-600. doi: 10.1016/j.biopsych.2010.10.023. Epub 2010 Dec 31. PMID 21195389
- [Background] Pearson NJ, Johnson LL, Nahin RL. Insomnia, trouble sleeping, and complementary and alternative medicine: Analysis of the 2002 national health interview survey data. Arch Intern Med. 2006 Sep 18;166(16):1775-82. doi: 10.1001/archinte.166.16.1775. PMID 16983058
- [Background] Castro LS, Poyares D, Leger D, Bittencourt L, Tufik S. Objective prevalence of insomnia in the Sao Paulo, Brazil epidemiologic sleep study. Ann Neurol. 2013 Oct;74(4):537-46. doi: 10.1002/ana.23945. Epub 2013 Sep 16. PMID 23720241
- [Background] Javaheri S, Redline S. Insomnia and Risk of Cardiovascular Disease. Chest. 2017 Aug;152(2):435-444. doi: 10.1016/j.chest.2017.01.026. Epub 2017 Jan 30. PMID 28153671
- [Background] Fernandez-Mendoza J, Vgontzas AN, Liao D, Shaffer ML, Vela-Bueno A, Basta M, Bixler EO. Insomnia with objective short sleep duration and incident hypertension: the Penn State Cohort. Hypertension. 2012 Oct;60(4):929-35. doi: 10.1161/HYPERTENSIONAHA.112.193268. Epub 2012 Aug 14. PMID 22892811
- [Background] Vgontzas AN, Liao D, Bixler EO, Chrousos GP, Vela-Bueno A. Insomnia with objective short sleep duration is associated with a high risk for hypertension. Sleep. 2009 Apr;32(4):491-7. doi: 10.1093/sleep/32.4.491. PMID 19413143
- [Background] Suka M, Yoshida K, Sugimori H. Persistent insomnia is a predictor of hypertension in Japanese male workers. J Occup Health. 2003 Nov;45(6):344-50. doi: 10.1539/joh.45.344. PMID 14676413
- [Background] Laugsand LE, Vatten LJ, Platou C, Janszky I. Insomnia and the risk of acute myocardial infarction: a population study. Circulation. 2011 Nov 8;124(19):2073-81. doi: 10.1161/CIRCULATIONAHA.111.025858. Epub 2011 Oct 24. PMID 22025601
- [Background] Mallon L, Broman JE, Hetta J. Sleep complaints predict coronary artery disease mortality in males: a 12-year follow-up study of a middle-aged Swedish population. J Intern Med. 2002 Mar;251(3):207-16. doi: 10.1046/j.1365-2796.2002.00941.x. PMID 11886479
- [Background] Laugsand LE, Strand LB, Platou C, Vatten LJ, Janszky I. Insomnia and the risk of incident heart failure: a population study. Eur Heart J. 2014 Jun 1;35(21):1382-93. doi: 10.1093/eurheartj/eht019. Epub 2013 Mar 5. PMID 23462728
- [Background] Han X, Yang Y, Chen Y, Gao L, Yin X, Li H, Qiu J, Wang Y, Zhou Y, Xia Y. Association between insomnia and atrial fibrillation in a Chinese population: A cross-sectional study. Clin Cardiol. 2017 Sep;40(9):765-769. doi: 10.1002/clc.22731. Epub 2017 May 31. PMID 28561943
- [Background] Li Y, Zhang X, Winkelman JW, Redline S, Hu FB, Stampfer M, Ma J, Gao X. Association between insomnia symptoms and mortality: a prospective study of U.S. men. Circulation. 2014 Feb 18;129(7):737-46. doi: 10.1161/CIRCULATIONAHA.113.004500. Epub 2013 Nov 13. PMID 24226807
- [Background] McGrath ER, Espie CA, Power A, Murphy AW, Newell J, Kelly C, Duffy N, Gunning P, Gibson I, Bostock S, O'Donnell MJ. Sleep to Lower Elevated Blood Pressure: A Randomized Controlled Trial (SLEPT). Am J Hypertens. 2017 Mar 1;30(3):319-327. doi: 10.1093/ajh/hpw132. PMID 28391289
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Marti-Soler H, Hirotsu C, Marques-Vidal P, Vollenweider P, Waeber G, Preisig M, Tafti M, Tufik SB, Bittencourt L, Tufik S, Haba-Rubio J, Heinzer R. The NoSAS score for screening of sleep-disordered breathing: a derivation and validation study. Lancet Respir Med. 2016 Sep;4(9):742-748. doi: 10.1016/S2213-2600(16)30075-3. Epub 2016 Jun 16. PMID 27321086
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- [Background] Chowdhuri S, Quan SF, Almeida F, Ayappa I, Batool-Anwar S, Budhiraja R, Cruse PE, Drager LF, Griss B, Marshall N, Patel SR, Patil S, Knight SL, Rowley JA, Slyman A; ATS Ad Hoc Committee on Mild Obstructive Sleep Apnea. An Official American Thoracic Society Research Statement: Impact of Mild Obstructive Sleep Apnea in Adults. Am J Respir Crit Care Med. 2016 May 1;193(9):e37-54. doi: 10.1164/rccm.201602-0361ST. PMID 27128710
- [Result] Edinger JD, Bonnet MH, Bootzin RR, Doghramji K, Dorsey CM, Espie CA, Jamieson AO, McCall WV, Morin CM, Stepanski EJ; American Academy of Sleep Medicine Work Group. Derivation of research diagnostic criteria for insomnia: report of an American Academy of Sleep Medicine Work Group. Sleep. 2004 Dec 15;27(8):1567-96. doi: 10.1093/sleep/27.8.1567. PMID 15683149